CLINICAL TRIAL: NCT01122095
Title: Cross-sectional Evaluation of Biological Markers of Cardiovascular Disease in Children and Adolescents With Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: Amgen (Industry)
Responsible Party: Lawrence Eichenfield, University of California, San Diego
Other Study IDs: 20080414
Record Dates: First submitted 2010-04-27; First posted 2010-05-12 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-04

CONDITIONS: Psoriasis; Obesity; Cardiovascular Risk; Inflammation
Keywords: Psoriasis; Cardiovascular risk
MeSH Terms: conditions — Psoriasis; Obesity; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Psoriasis: Children with psoriasis Age matched controls without psoriasis or other significant inflammatory disease
- Control patient: Age matched, without psoriasis or significant inflammatory disease

SUMMARY:
Hypothesis 1: Patients with psoriasis will have clinical and laboratory assessments differing from control patients.

Hypothesis 2: Patients with psoriasis will have laboratory alterations that correlate with other clinical characteristics of their psoriasis.

DETAILED DESCRIPTION:
Psoriasis was initially considered an inflammatory condition primarily of the skin. However, advances in medical knowledge have allowed insight into the wide-ranging systemic effects of long-term uncontrolled inflammation, thus shifting the concept of psoriasis from an inflammatory disease restricted to the skin to a systemic process. Adults w/ psoriasis have higher rates of obesity, hypertension, diabetes, hyperlipidemia and smoking and the prevalence of each risk factor increases as the extent of psoriasis increases.1 It is uncertain if any of this relates to a behavioral reaction to having psoriasis or as a separate part of the disease process. Inflammation has a role in the pathogenesis of cardiovascular disease most noted by multiple observational studies of psoriasis patients which demonstrate an increased risk of arterial or venous events, notably myocardial infarction, cerebrovascular events, pulmonary emboli, cardiovascular death or mortality overall. Specifically, Gelfand et. al. show an increased relative risk for myocardial infarction and an increased hazard ratio for mortality in patients with severe psoriasis, but most notably, show highest risk in younger adult patients. There is a paucity of data on risks with psoriasis in the pediatric and adolescent age group.

ELIGIBILITY:
Inclusion Criteria:

Subjects of any race or ethnicity who meet all of the following criteria are eligible for enrollment into the study:

1. The subject has a diagnosis of typical psoriasis, with or without arthritis, based on the clinical evaluation by an investigator or a prior diagnosis by a pediatric dermatologist
2. Persons residing in the US.
3. Subjects 0 to 18 years of age.
4. Subjects/Guardians willing and able to comply with the requirements of the study.
5. Subjects/Guardians willing and able to give informed consent.
6. The subject is in general good health in the opinion of the investigator.

Exclusion Criteria:

1. Over 18 years of age.
2. Subject has had a diagnosis of congenital heart disease.
3. Subject has had any cardiac catheterizations or surgeries.
4. Subject has taken any cardiac medications (calcium channel blockers, beta blockers, vasotropic medicines) within the past 2 years.
5. Subjects determined to have atypical psoriasis or isolated palmoplantar psoriasis.
6. Subject diagnosed with any other systemic inflammatory disease including atopic dermatitis, severe acne vulgaris, inflammatory bowel disease, juvenile idiopathic arthritis, connective tissue disease and other similar conditions.
7. Having autoimmune or immunodeficiency disease.
8. Presence of active systemic fungal, bacterial, or viral infections.
9. Presence of active systemic malignancy.
10. Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
11. Inability or unwillingness of a participant to give written informed consent.

Control Inclusion Criteria:

1. Age up to 18 years.
2. Ability and willingness to provide informed consent.

Control Exclusion Criteria:

1. Over 18 years of age.
2. Subject has had a diagnosis of congenital heart disease.
3. Subject has had any cardiac catheterizations or surgeries.
4. Subject has taken any cardiac medications (calcium channel blockers, beta blockers, vasotropic medicines) within the past 2 years.
5. Subjects determined to have psoriasis of any type or a family history (first degree relative) with psoriasis.
6. Subject diagnosed with any other systemic inflammatory disease including atopic dermatitis, severe acne vulgaris, inflammatory bowel disease, juvenile idiopathic arthritis, connective tissue disease and other similar conditions.
7. Having autoimmune or immunodeficiency disease.
8. Presence of active systemic fungal, bacterial, or viral infections.
9. Presence of active systemic malignancy.
10. Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements.
11. Inability or unwillingness of a participant to give written informed consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: case subjects, male or female, with typical psoriasis, with or without arthritis, ages 0 to 18 years of age and of all races and ethnicities control subjects, male or female, normal, health, non-soriatic subjects, 0 to 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Obesity risk assessment | 6 months
  Body Mass Index; C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence F. Eichenfield, MD, Principal Investigator — University of Calfornia, San Diego
Locations (1):
- Rady Children's Hospital Dermatolgoy, San Diego, California, United States

REFERENCES:
- [Background] 1. Neimann AL, Shin DB, Wang X, Margolis DJ, Troxel AB , Gelfand JM. Prevalence of cardiovascular risk factors in patients with psoriasis. J Am Acad Dermatol 2006;55:829-35. 2. Gelfand J, Neimann A, Shin D et al. Risk of myocardial infarction in patients with psoriasis. JAMA. 2006;296:1735-1741. 3. Gelfand J, Troxel B, Lewis J et al. The risk of mortality in patients with psoriasis: Results from a population-based study. Arch Dermatol. 2007;143(12):1493-1499 4. Kelishadi R, Ardalan G, Gheiratmand R, Adeli K, Delavari A, and Majdzadeh R et al. Pediatric metabolic syndrome and associated anthropometric indices: the CASPIAN study. Acta Paediatrica, 2006. 95: 1625-1634. 5. Goodman E, Dolan L, Morrison J and Daniels S. Factor Analysis of Clustered Cardiovascular Risks in Adolescence. Circulation 2005; 111: 1970-1977. 6. Schwimmer JB, Pardee PE, Lavine JE, Blumkin AK, Cook S. Cardiovascular Risk Factors and the Metabolic Syndrome in Pediatric Nonalcoholic Fatty Liver Disease. Circulation. 2008 June. 118:277-283.